CLINICAL TRIAL: NCT00044356
Title: A Phase II Study of High-Dose Allovectin-7® in Patients With Advanced Metastatic Melanoma
Brief Title: Phase II Trial of Allovectin-7® for Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vical (Industry)
Responsible Party: Dmitri D. Kharkevitch, MD, PhD, Vical Incorporated
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VCL-1005-208; NCT00028444 (obsolete NCT alias)
Record Dates: First submitted 2002-08-26; First posted 2002-08-28 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Melanoma; Metastatic Melanoma; Malignant Melanoma; Skin Cancer
Keywords: Melanoma; Metastatic Melanoma; Malignant Melanoma; Skin Cancer; Tumor; Experimental Treatment; Clinical Trial; Gene Therapy; Gene Delivery; Gene Transfer; Immunotherapy; Cancer; Neoplasm; Lesion; Metastasis; Cancerous mole; Melanoma vaccine; Cancer research; Cancer cells; Allovectin-7®
MeSH Terms: conditions — Melanoma; Skin Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Allovectin-7

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: Allovectin-7®

SUMMARY:
The purpose of this clinical trial is to determine if Allovectin-7®, an experimental gene-based immunotherapy, can shrink melanoma tumors. The trial will also examine if this treatment can improve the time to disease progression.

DETAILED DESCRIPTION:
Treatment - If you take part in this trial you will be treated for about 10 weeks. You will receive an injection of Allovectin-7® by needle, directly into one or more selected tumors once a week for the first six weeks. The injections may be given in a doctor's office. During a four-week observation period, your disease will be measured to see if the treatment is working. This will be done by general physical exams and scans (such as X-ray scans). Patients who show no sign of disease progression may be offered an option to repeat this treatment course.

ELIGIBILITY:
In order to be in this trial, you must meet the enrollment criteria. Below is a list of some of the enrollment criteria.

* You have been diagnosed with Stage III or Stage IV melanoma
* Your cancer has returned after a prior treatment (e.g. radiation or chemotherapy) or you refused therapy with standard treatment
* You are able to carry out your normal daily activities
* Your melanoma has not spread to your brain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2001-02; Primary Completion 2004-08 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas Cancer Research Center, Little Rock, Arkansas
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Louisiana State University Medical Center, New Orleans, Louisiana
  - Hematology Oncology Associates of Baltimore, Baltimore, Maryland
  - North Memorial Health Care, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - The Melanoma Center of Saint Louis, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Beth Israel Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - Cancer Care Alliance, Seattle, Washington